CLINICAL TRIAL: NCT04356040
Title: Safety and Effectiveness of the TactiFlex(TM) Ablation Catheter, Sensor Enabled(TM) (TactiFlex SE) for Treating Drug-refractory, Symptomatic Atrial Fibrillation.
Brief Title: TactiFlex Paroxysmal Atrial Fibrillation IDE Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10303; CRD_978 (Other: Abbott)
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a prospective non-randomized parallel-assignment multi-center clinical investigation. The study design includes two subject cohorts: 1) Paroxysmal Atrial Fibrillation Main Study, and 2) Paroxysmal Atrial Fibrillation High Standard Power Substudy. Subjects in the main study cohorts are to be treated using the full range of ablation power settings in the Instructions For Use. Subjects in the Substudy are to be treated in the upper end of the recommended ablation power settings (40-50 Watts).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Main Study (Experimental)
  Interventions: Device: TactiFlex SE
- High Standard Power Sub-Study (Experimental)
  Interventions: Device: TactiFlex SE - High Standard Power

INTERVENTIONS:
Device: TactiFlex SE — Radiofrequency ablation with the TactiFlex SE ablation catheter. The procedure should be performed according to the TactiFlex SE investigational Instructions for Use document using the recommended ablation parameters as noted in the document.
  Other Names: TactiFlex Sensor Enabled Ablation Catheter
  Arms: Main Study
Device: TactiFlex SE - High Standard Power — Radiofrequency ablation with the TactiFlex SE ablation catheter. Subjects in the High Standard Power Substudy are to undergo the same study procedures as subjects in the main study, except that ablation power settings of 40-50 Watts are to be used in the left atrium, unless there is a medical reason to use a lower power.
  Arms: High Standard Power Sub-Study

SUMMARY:
Prospective non-randomized parallel-assignment multi-center clinical investigation. The study design includes two subject cohorts: 1) Paroxysmal Atrial Fibrillation Main Study, and 2) Paroxysmal Atrial Fibrillation High Standard Power Substudy. Subjects in the main study cohorts are to be treated using the full range of ablation power settings in the Instructions For Use. Subjects in the High Standard Power Substudy are to be treated in the upper end of the recommended ablation power settings (40-50 Watts).

DETAILED DESCRIPTION:
This clinical investigation is intended to demonstrate the safety and effectiveness of the TactiFlex(TM) Ablation Catheter, Sensor Enabled(TM) (TactiFlex SE) for treating drug-refractory, symptomatic paroxysmal atrial fibrillation. This clinical investigation will be conducted under an investigational device exemption and is intended to support market approval of the TactiFlex SE catheter worldwide. Three hundred and Fifty Five (355) subjects will be enrolled at up to 50 investigational sites worldwide. This clinical investigation is sponsored by Abbott.

ELIGIBILITY:
A patient will be eligible for clinical trial participation if he/she meets the following criteria:

1. Plans to undergo a catheter ablation procedure due to symptomatic paroxysmal atrial fibrillation
2. Physician's note indicating recurrent self-terminating atrial fibrillation
3. One electrocardiographically documented atrial fibrillation episode within 12-months prior to informed consent/enrollment. Documented evidence of the atrial fibrillation episode must either be continuous atrial fibrillation on a 12-lead ECG or include at least 30 seconds of atrial fibrillation from another ECG device.
4. At least 18 years of age
5. Able and willing to comply with all trial requirements
6. Informed of the nature of the trial, agreed to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical trial site.

A patient will be excluded from enrollment in the clinical trial if he/she meets any of the following criteria:

1. Persistent or long-standing persistent atrial fibrillation
2. Active systemic infection
3. Known presence of cardiac thrombus
4. Hypertrophic cardiomyopathy
5. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, and other major surgical procedures in the 90-day period preceding procedure
6. Myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, or valve or coronary bypass grafting surgery within 90 days of procedure
7. Left atrial diameter > 5.0 cm measured within 180 days of procedure (echocardiography or computerized tomography)
8. Left ventricular ejection fraction < 35% measured within 180 days of procedure (echocardiography or computerized tomography)
9. New York Heart Association class III or IV
10. Previous left atrial surgical or catheter ablation procedure
11. Left atrial surgical procedure or incision with resulting scar (including left atrial appendage closure device)
12. Previous tricuspid or mitral valve replacement or repair
13. Heart disease in which corrective surgery is anticipated within 180 days after the procedure
14. Bleeding diathesis or suspected pro-coagulant state
15. Contraindication to long term anti-thromboembolic therapy
16. Presence of any condition that precludes appropriate vascular access
17. Renal failure requiring dialysis
18. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
19. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
20. Women who are pregnant or breastfeeding
21. Presence of other anatomic or comorbid condition that, in the investigator's opinion, could limit the patient's ability to participate in the clinical trial or to comply with follow up requirements, or impact the scientific soundness of the clinical trial results
22. Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this clinical trial
23. Patient is unlikely to survive the protocol follow up period of 12-months after the procedure
24. Body mass index > 40 kg/m2
25. Presence of other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
26. Individuals without legal authority
27. Individuals unable to read or write
28. Patients who have had a ventriculotomy or atriotomy within the preceding 4 weeks of procedure,
29. Patients with prosthetic valves,
30. Patients with a myxoma,
31. Patients with an interatrial baffle or patch as the transseptal puncture could persist and produce an iatrogenic atrial shunt
32. Patient unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
33. Stroke or transient ischemic attack within the last 90 days
34. Stent, constriction, or stenosis in a pulmonary vein.
35. Rheumatic heart disease
36. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ruffner, PhD, Study Director — Clinical Program Director
Locations (45):
- United States (30):
  - Affinity Cardiovascular Specialists, LLC, Birmingham, Alabama
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Mills-Peninsula Medical Center, Burlingame, California
  - Scripps Health, La Jolla, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Kootenai Heart Clinics, Coeur d'Alene, Idaho
  - St. Vincent Hospital, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Providence Hospital, Southfield, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - New York University Hospital, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Franciscan Heart & Vascular Associates, Tacoma, Washington
- Australia (5):
  - Westmead Hospital, Westmead, New South Wales
  - Wesley Private Hospital, Auchenflower, Queensl
  - The Prince Charles Hospital, Chermside, Queensl
  - Monash Medical Centre, Clayton, Victori
  - Royal Adelaide Hospital, Adelaide
- A. ö. Krankenhaus der Elisabethinen Linz, Linz, UPR AUS, Austria
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- IKEM Prague, Prague, Cbohmia, Czechia
- Germany (2):
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen, N. RHIN
  - Herzzentrum Leipzig GmbH, Leipzig
- Prince of Wales Hospital, Hong Kong, HONG KO, Hong Kong
- Ospedale San Raffaele, Milan, Lombard, Italy
- Erasmus MC - Thoraxcenter, Rotterdam, S Holln, Netherlands
- Taipei Veterans General Hospital (VGH), Taipei, Ntaiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxysmal AF - Main Study: TactiFlex SE: Radiofrequency ablation with the TactiFlex SE ablation catheter. The procedure should be performed according to the TactiFlex SE investigational Instructions for Use document using the recommended ablation parameters as noted in the document.
- Paroxysmal AF HSP Sub-Study: TactiFlex SE - HSP: Radiofrequency ablation with the TactiFlex SE ablation catheter. Subjects in the HSP Substudy are to undergo the same study procedures as subjects in the main study, except that ablation power settings of 40-50 Watts are to be used in the left atrium, unless there is a medical reason to use a lower power.
Period: Overall Study
Arm/Group | Paroxysmal AF - Main Study | Paroxysmal AF HSP Sub-Study
Started | 305 | 50
Device Inserted and RF Energy Delivered | 284 | 50
7-Day Visit | 280 | 50
5-Week Visit | 279 | 50
3-Month Visit | 272 | 50
6-Month Visit | 267 | 49
12-Month Visit | 264 | 48
Completed | 268 | 48
Not Completed | 37 | 2
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 13 | 1
Not completed — Enrollment Pause | 10 | 0
Not completed — Did not meet Inclusion/Exclusion criteria | 7 | 0
Not completed — Procedure aborted prior to device insertion into the vasculature | 1 | 0
Not completed — PI left institution | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxysmal AF - Main Study | Paroxysmal AF HSP Sub-Study | Total
Number analyzed (Participants) | 284 | 50 | 334
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.0 [56.0 to 71.0] | 67.0 [61.0 to 70.0] | 65.0 [56.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 16 | 120
  Male | 180 | 34 | 214
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 264 | 45 | 309
  Unknown or Not Reported | 15 | 3 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 262 | 44 | 306
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 3
  Austria | 29 | 0 | 29
  Hong Kong | 3 | 0 | 3
  United States | 185 | 50 | 235
  Czechia | 7 | 0 | 7
  Taiwan | 2 | 0 | 2
  Italy | 2 | 0 | 2
  Australia | 31 | 0 | 31
  Germany | 22 | 0 | 22
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.4 [25.6 to 33] | 28.35 [25.9 to 30.4] | 28.4 [25.7 to 32.8]
CHA2DS2Vasc Score [Median (Inter-Quartile Range); unit: units on a scale] — This scoring system includes the following risk factors
  C for Congestive heart failure adds 1 point. H for Hypertension or high blood pressure adds 1 point A for Age greater than or equal to 75 years adds 2 points D for Diabetes mellitus or type 2 diabetes adds 1 point S for prior Stroke or TIA adds 2 points V for Vascular disease adds 1 point A for Age between 65 and 74 years adds 1 point S for female Sex adds 1 point
  Range 0-9. A higher score is considered at higher risk for stroke.
  Note: while the points above add to 10, you can only have a max of 2 points for age.
  units on a scale | 2 [1.0 to 3.0] | 2 [2.0 to 3.0] | 2 [2.0 to 3.0]
New York Heart Association Functional Classification [Count of Participants; unit: Participants] — The New York Heart Association Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  Class I = no limitation of physical activity. Class II = slight limitation Class III = marked limitation Class IV = unable to carry on any physical activity without discomfort
  Participants
    No Heart Failure | 203 | 44 | 247
    Class I | 54 | 1 | 55
    Class II | 27 | 5 | 32
    Class III or IV | 0 | 0 | 0
Left Ventricular Ejection Fraction [Median (Inter-Quartile Range); unit: Percentage] — Percentage of left ventricular ejection as determined using an echo or computerized tomography scan.
  Percentage | 60.0 [55.0 to 60.0] | 55.0 [55.0 to 60.0] | 60.0 [55.0 to 60.0]
Left Atrial Diameter [Median (Inter-Quartile Range); unit: Millimeters] — As measured by an echo or computerized tomography scan.
  Millimeters | 40.0 [36.0 to 43.0] | 40.0 [36.0 to 43.0] | 40.0 [36.0 to 43.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device or Procedure-related Serious Adverse Events
Description: Tthe rate of device and/or procedure-related serious adverse events with onset within 7-days of any ablation procedure that uses the TactiFlex SE catheter (initial or repeat procedure performed 31-80 days of initial procedure) that are defined below:
  * Atrio-esophageal fistula1
  * Cardiac tamponade/perforation1
  * Death
  * Heart block
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve injury resulting in diaphragmatic paralysis
  * Pulmonary edema
  * Pulmonary vein stenosis1
  * Stroke/cerebrovascular accident
  * Thromboembolism
  * Transient ischemic attack
  * Vagal nerve injury/gastroparesis
  * Vascular access complications (including major bleeding events)
    1. Atrio-esophageal fistula, cardiac tamponade/perforation and pulmonary vein stenosis will be evaluated through 12-months.
Time Frame: Through 12 months
Population: The primary safety analysis population for the primary safety endpoint included all treated subjects who have completed their 7-day follow-up visit; or crossed the end of the 7-day visit window without the visit but with a primary safety endpoint event.
Measure: Count of Participants; unit: Participants
Arm/Group | Main Study | High Standard Power Sub-Study
Number analyzed (Participants) | 280 | 50
Participants | 12 | 2

2. Primary Outcome: KM Rate of Freedom From Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia Recurrence
Description: Freedom from documented (symptomatic or asymptomatic) Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia episodes of >30 seconds duration that are documented by 12-lead ECG, transtelephonic monitoring or Holter monitor after the initial catheter ablation procedure through 12-months of follow-up. Recurrence during the 90-day blanking period will not be considered a treatment failure. One repeat procedure will be allowed during the blanking period. Failure to achieve acute procedural success during the last ablation procedure with the TactiFlex SE catheter will constitute failure. After the 90-day blanking period, use of Class I or III anti-arrhythmic drugs will not count as a therapy failure provided that only previously failed drugs are taken at doses that do not exceed the previously failed dose.
Time Frame: Through 12 months
Population: All treated subjects
Measure: Number (97.5% Confidence Interval); unit: percentage
Arm/Group | Main Study | High Standard Power Sub-Study
Number analyzed (Participants) | 284 | 50
percentage | 72.9 [67.2 to 78.6] | 71.8 [57.0 to 86.6]

3. Secondary Outcome: KM Rate of Freedom From Symptomatic Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia Recurrence
Description: Freedom from documented symptomatic atrial fibrillation/atrial flutter/atrial tachycardia episodes of >30 seconds duration that are documented by 12-lead ECG, transtelephonic monitoring or Holter monitor after the initial catheter ablation procedure through 12-months of follow-up. Recurrence during the 90-day blanking period (≤90 days post-initial procedure) will not be considered a treatment failure. One repeat procedure will be allowed for ablation 31-80 days after the initial procedure and will not be considered a treatment failure. Failure to achieve acute procedural success during the last ablation procedure with the TactiFlex SE catheter will constitute failure. After the 90-day blanking period, use of Class I or III anti-arrhythmias drugs will not count as a therapy failure provided that only previously failed Class I or III anti-arrhythmias drugs are taken at doses that do not exceed the previously failed dose.
Time Frame: Through 12 months
Population: All Treated Subjects
Measure: Number (97.5% Confidence Interval); unit: percentage
Arm/Group | Main Study | High Standard Power Sub-Study
Number analyzed (Participants) | 284 | 50
percentage | 80.4 [75.2 to 85.6] | 75.9 [61.5 to 90.3]

4. Secondary Outcome: KM Rate of Freedom From Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia Recurrence With Only 1 Ablation Procedure
Description: Freedom from documented (symptomatic or asymptomatic) Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia episodes of >30 seconds duration that are documented by 12-lead ECG, transtelephonic monitoring or Holter monitor after the initial catheter ablation procedure through 12-months of follow-up. Recurrence during the 90-day blanking period (≤90 days post-initial procedure) will not be considered a treatment failure. Any repeat ablation procedure in the left atrium will be considered a treatment failure. Failure to achieve acute procedural success during the ablation procedure with the TactiFlex SE catheter will constitute failure. After the 90-day blanking period, use of Class I or III anti-arrhythmic drugs will not count as a therapy failure provided that only previously failed Class I or III anti-arrhythmic drugs are taken at doses that do not exceed the previously failed dose.
Time Frame: 12 months
Population: All treated subjects
Measure: Number (97.5% Confidence Interval); unit: percentage
Arm/Group | Main Study | High Standard Power Sub-Study
Number analyzed (Participants) | 284 | 50
percentage | 71.5 [65.7 to 77.3] | 71.8 [57.0 to 86.6]

5. Secondary Outcome: KM Rate of Freedom From Atrial Fibrillation, Atrial Flutter or Atrial Tachycardia Recurrence, Without Anti-arrhythmic Drugs
Description: Freedom from documented (symptomatic or asymptomatic) Atrial Fibrillation/Atrial Flutter/Atrial Tachycardia episodes of >30 seconds duration that are documented by 12-lead ECG, transtelephonic monitoring or Holter monitor after the initial catheter ablation procedure through 12-months of follow-up (9 months after a 90-day blanking period). Recurrence during the 90-day blanking period (≤90 days post-initial procedure) will not be considered a treatment failure. One repeat procedure will be allowed for ablation 31-80 days after the initial procedure and will not be considered a treatment failure. Failure to achieve acute procedural success during the last ablation procedure with the TactiFlex SE catheter will constitute failure. After the 90-day blanking period, any use of a Class I or III anti-arrhythmic drugs will count as an effectiveness failure.
Time Frame: Through 12 months
Population: All treated subjects
Measure: Number (97.5% Confidence Interval); unit: percentage
Arm/Group | Main Study | High Standard Power Sub-Study
Number analyzed (Participants) | 284 | 50
percentage | 64.0 [58.0 to 70.0] | 65.8 [50.9 to 80.7]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Paroxysmal AF - Main Study | Paroxysmal AF HSP Sub-Study
All-Cause Mortality (participants affected / at risk) | 2/284 | 0/50
Serious Adverse Events (participants affected / at risk) | 65/284 | 8/50
Other Adverse Events (participants affected / at risk) | 5/284 | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxysmal AF - Main Study (N=284) | Paroxysmal AF HSP Sub-Study (N=50)
Infection (Infections and infestations) | 9 (10) | 2 (2)
Arrhythmia Pre-Existing (Cardiac disorders) | 8 (8) | 0 (0)
Cancer/Non-Malignant Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 4 (4) | 0 (0)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Chest Pain/Angina (Cardiac) (Cardiac disorders) | 3 (3) | 0 (0)
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Vascular Access Complications (Vascular disorders) | 3 (3) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 2 (2) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 2 (2) | 1 (1)
Pain (Non-Cardiac) (General disorders) | 2 (2) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 0 (0)
Syncope/Dizziness (General disorders) | 2 (2) | 0 (0)
Thrombosis/Thrombus (Cardiac disorders) | 1 (2) | 0 (0)
Vascular Bleeding/Local Hematomas Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Abnormal Labs (e.g., Creatine phosphokinase, Creatinine, Troponin) (General disorders) | 1 (1) | 0 (0)
Arrhythmia New (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block/Bundle Branch Block (Cardiac disorders) | 1 (1) | 0 (0)
Bleeding/Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac Perforation/Injury (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident/Stroke (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Endocrine Disease/Disorder (Endocrine disorders) | 1 (1) | 0 (0)
Heart Failure/Pump Failure (Cardiac disorders) | 1 (1) | 0 (0)
Nerve System Damage/Injury/Disease (Nervous system disorders) | 1 (1) | 0 (0)
Renal Decompensation/Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Valvular Damage or Insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Vascular Damage (e.g., Perforation, Dissection, Obstruction) (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vasovagal Reaction (General disorders) | 1 (1) | 0 (0)
Volume Overload (General disorders) | 1 (1) | 0 (0)
Abnormal Vision (Eye disorders) | 0 (0) | 1 (1)
Elective Procedure/Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Other: Diarrhea (General disorders) | 0 (0) | 1 (1)
Other: Urinary/Urine Retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Other: Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Other: Aortic Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Other: Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Other: Collapsed Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other: Motorcycle Crash (General disorders) | 1 (1) | 0 (0)
Other: Pericardial-Esophageal Fistula (Cardiac disorders) | 1 (1) | 0 (0)
Other: Pseudoaneurysm of Common Femoral Artery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other: Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other: Spontaneous Subarachnoid Hemorrhage (General disorders) | 1 (1) | 0 (0)
Other: Ureteral Calculus/Stone (Renal and urinary disorders) | 2 (2) | 0 (0)
Other: Urinary Frequency Needing transurethral resection of the prostate (Renal and urinary disorders) | 1 (1) | 0 (0)
Other: Urinary Retention with Acute Kidney Injury (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxysmal AF - Main Study (N=284) | Paroxysmal AF HSP Sub-Study (N=50)
Volume Overload (Endocrine disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data and results from the clinical investigation are the sole property of the Sponsor. The Investigators will not use this clinical investigation-related data without the written consent of the Sponsor for any purpose other than for clinical investigation completion or for generation of publication materials, as referenced in the Clinical Trial Agreement. Single-center results are not allowed to be published or presented before the multi-center results.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT04356040/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04356040/SAP_002.pdf